CLINICAL TRIAL: NCT05539976
Title: An Open-label Taste Assessment of Iberdomide and Mezigdomide in Healthy Participants
Brief Title: A Taste Assessment of Iberdomide and Mezigdomide in Healthy Participants
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM048-015
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy participants who perform taste evaluations: A maximum of 10 healthy adult participants will complete a maximum of 30 taste assessment days, to evaluate the taste characteristics of iberdomide or mezigdomide on each taste assessment day.

SUMMARY:
The purpose of this study is to develop taste profiles of iberdomide and mezigdomide drug substances and oral formulation prototypes in order to develop a pediatric oral form of iberdomide and mezigdomide.

ELIGIBILITY:
Inclusion Criteria:

* Participant is qualified based on training and experience.
* Participants must be trained to detect, identify, recognize, and accurately describe different taste elements and flavor combinations. Training is initially accomplished by tasting model compounds and learning to recognize and describe these accurately. These abilities are then honed and refined through additional experience in performing taste profiling.
* Participant is qualified based on training and experience.
* Senopsys LLC will provide all participants.
* Participants must be trained to detect, identify, recognize, and accurately describe different taste elements and flavor combinations. Training is initially accomplished by tasting model compounds and learning to recognize and describe these accurately. These abilities are then honed and refined through additional experience in performing taste profiling.

Exclusion Criteria:

* Participant has any history of any illness, medical condition, laboratory abnormality, or psychiatric illness that, in the opinion of the investigator, might confound the results of the study or places the participant at unacceptable risk if he or she were to participate in the study.
* Participant has a known hypersensitivity to mezigdomide, iberdomide, thalidomide, lenalidomide, or pomalidomide.
* Participant is a female that is pregnant, breastfeeding, or is a women of childbearing potential (WOCBP).

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of healthy volunteers who are qualified based on training and experience in performing taste evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Taste Evaluation - Aromatic Identity | Up to 3 Months
Taste Evaluation - Amplitude | Up to 3 Months
Taste Evaluation - Mouthfeel | Up to 3 Months
Taste Evaluation - Off-notes | Up to 3 Months
Taste Evaluation - Aftertaste | Up to 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Woburn, Massachusetts, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm